CLINICAL TRIAL: NCT03179436
Title: A Phase 1 / 2 Open Label, Multi-Arm, Multicenter Study of MK-1308 in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: Study of Quavonlimab (MK-1308) in Combination With Pembrolizumab (MK-3475) in Advanced Solid Tumors (MK-1308-001)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1308-001; MK-1308-001 (Other: Merck); 173820 (Registry Identifier: JAPIC-CTI); 2019-003703-35 (EudraCT Number)
Record Dates: First submitted 2017-05-31; First posted 2017-06-07 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors
Keywords: Programmed Cell Death Protein 1 (PD-1, PD1),; Programmed Cell Death Ligand 1 (PD-L1, PDL1); Programmed Cell Death Ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Escalation: Dose Level (DL) 1 Quavonlimab + Pembro: Cohort 1 (Experimental): On Cycle 1, Day 1 of the Dose Escalation Phase, advanced solid tumor participants receive a single monotherapy dose lead-in with quavonlimab at dose level 1 (DL1). On Cycle 2, Day 1, and for 3 subsequent cycles on Day 1 (Cycles 3 to 5), these participants receive quavonlimab at DL1 in combination with pembrolizumab (pembro) at pembrolizumab dose level 1 (PDL1) according to Schedule 1. For all subsequent cycles (starting with Cycle 6), all participants receive pembrolizumab monotherapy according to Schedule 1. Participants will be treated for up to 35 cycles total on study.
  Interventions: Biological: Quavonlimab; Biological: Pembrolizumab
- Escalation: DL 2 Quavonlimab + Pembro: Cohort 2 (Experimental): On Cycle 1, Day 1 of the Dose Escalation Phase, participants with advanced solid tumors except NSCLC receive a single monotherapy dose lead-in with quavonlimab at DL2. On Cycle 2, Day 1, and for 3 subsequent cycles on Day 1 (Cycles 3 to 5), these participants receive quavonlimab at DL2 in combination with pembrolizumab at PDL1 according to Schedule 1. For all subsequent cycles (starting with Cycle 6), all participants receive pembrolizumab monotherapy according to Schedule 1. Participants will be treated for up to 35 cycles total on study.
  Interventions: Biological: Quavonlimab; Biological: Pembrolizumab
- Escalation: DL 3 Quavonlimab + Pembro: Cohort 3 (Experimental): On Cycle 1, Day 1 of the Dose Escalation Phase, participants with advanced solid tumors except NSCLC receive a single monotherapy dose lead-in with quavonlimab at DL3. On Cycle 2, Day 1, and for 3 subsequent cycles on Day 1 (Cycles 3 to 5), these participants receive quavonlimab at DL3 in combination with pembrolizumab at PDL1 according to Schedule 1. For all subsequent cycles (starting with Cycle 6), all participants receive pembrolizumab monotherapy according to Schedule 1. Participants will be treated for up to 35 cycles total on study.
  Interventions: Biological: Quavonlimab; Biological: Pembrolizumab
- Confirmation: DL 1 Quavonlimab Schedule 1 + Pembro (NSCLC): Arm A (Experimental): On Cycle 1, Day 1 of the Dose Confirmation Phase and during all subsequent cycles, participants with NSCLC receive quavonlimab at DL1 in combination with pembrolizumab at PDL1, both according to Schedule 1. Participants will be treated for up to 35 cycles total on study.
  Interventions: Biological: Quavonlimab; Biological: Pembrolizumab
- Confirmation: DL 1 Quavonlimab Schedule 2 + Pembro (NSCLC): Arm B (Experimental): On Cycle 1, Day 1 of the Dose Confirmation Phase, participants with NSCLC receive quavonlimab at DL1 in combination with pembrolizumab at PDL1. On all subsequent cycles, participants receive pembrolizumab at PDL1 according to Schedule 1 and quavonlimab at DL1 according to Schedule 2. Participants will be treated for up to 35 cycles total on study.
  Interventions: Biological: Quavonlimab; Biological: Pembrolizumab
- Confirmation: DL 2 Quavonlimab Schedule 2 + Pembro (NSCLC): Arm C (Experimental): On Cycle 1, Day 1 of the Dose Confirmation Phase, participants with NSCLC receive quavonlimab at DL2 in combination with pembrolizumab at PDL1. On all subsequent cycles, participants receive pembrolizumab at PDL1 according to Schedule 1 and at DL2 quavonlimab according to Schedule 2. Participants will be treated for up to 35 cycles total on study.
  Interventions: Biological: Quavonlimab; Biological: Pembrolizumab
- Confirmation: DL 2 Quavonlimab Schedule 2 + Pembro (SCLC): Arm D (Experimental): On Cycle 1, Day 1 of the Dose Confirmation Phase, participants with SCLC receive quavonlimab at DL2 in combination with pembrolizumab at PDL1. On all subsequent cycles, participants receive pembrolizumab at PDL1 according to Schedule 1 and quavonlimab at DL2 according to Schedule 2. Participants will be treated for up to 35 cycles total on study.
  Interventions: Biological: Quavonlimab; Biological: Pembrolizumab
- Confirmation: DL 2 Quavonlimab Schedule 1 + Pembro (NSCLC): Arm E (Experimental): On Cycle 1, Day 1 of the Dose Confirmation Phase and during all subsequent cycles, participants with NSCLC receive quavonlimab at DL2 in combination with pembrolizumab at PDL1 according to Schedule 1. Participants will be treated for up to 35 cycles total on study.
  Interventions: Biological: Quavonlimab; Biological: Pembrolizumab
- Expansion: DL1 Quavonlimab Schedule 2+PDL2 Pembro Schedule 2: Arm F (Experimental): On Cycle 1, Day 1 of the Efficacy Expansion Phase and during all subsequent cycles, participants with PD-1/PD-L1 refractory melanoma receive quavonlimab at DL1 in combination with pembrolizumab at pembrolizumab dose level 2 (PDL2). Both quavonlimab and pembrolizumab will be administered according to Schedule 2 for up to 24 months on study.
  Interventions: Biological: Quavonlimab; Biological: Pembrolizumab
- Expansion: DL1 Quavonlimab Schedule 2 Monotherapy: Arm G (Experimental): On Cycle 1, Day 1 of the Efficacy Expansion Phase and during all subsequent cycles, participants with PD-1/PD-L1 refractory melanoma receive quavonlimab at DL1 according to Schedule 2 for up to 24 months on study. Participants who demonstrate radiographically confirmed progressive disease in Arm G will be eligible to receive combination therapy with pembrolizumab (crossover).
  Interventions: Biological: Quavonlimab
- Coformulation: Pembrolizumab/Quavonlimab Schedule 2: Arm I (Experimental): On Cycle 1, Day 1 of the Coformulation Phase and during all subsequent cycles, participants with advanced/metastatic solid tumors receive pembrolizumab/quavonlimab according to Schedule 2 for up to 24 months on study.
  Interventions: Drug: Pembrolizumab/Quavonlimab
- Coformulation Phase in China: Pembrolizumab/Quavonlimab Schedule 2: Arm K (Experimental): On Cycle 1, Day 1 of the Coformulation Phase and during all subsequent cycles, participants in mainland China with advanced solid tumors receive pembrolizumab/quavonlimab according to Schedule 2 for up to 24 months on study.
  Interventions: Drug: Pembrolizumab/Quavonlimab

INTERVENTIONS:
Biological: Quavonlimab — Quavonlimab is administered intravenously (IV) during the Dose Escalation Phase and Dose Confirmation Phase at either DL1 or DL2, and is administered IV during the Efficacy Expansion Phase at DL2.
  Other Names: MK-1308
  Arms: Confirmation: DL 1 Quavonlimab Schedule 1 + Pembro (NSCLC): Arm A; Confirmation: DL 1 Quavonlimab Schedule 2 + Pembro (NSCLC): Arm B; Confirmation: DL 2 Quavonlimab Schedule 1 + Pembro (NSCLC): Arm E; Confirmation: DL 2 Quavonlimab Schedule 2 + Pembro (NSCLC): Arm C; Confirmation: DL 2 Quavonlimab Schedule 2 + Pembro (SCLC): Arm D; Escalation: DL 2 Quavonlimab + Pembro: Cohort 2; Escalation: DL 3 Quavonlimab + Pembro: Cohort 3; Escalation: Dose Level (DL) 1 Quavonlimab + Pembro: Cohort 1; Expansion: DL1 Quavonlimab Schedule 2 Monotherapy: Arm G; Expansion: DL1 Quavonlimab Schedule 2+PDL2 Pembro Schedule 2: Arm F
Biological: Pembrolizumab — Pembrolizumab is administered IV at PDL1 on Day 1 of each cycle starting Cycle 2 for the Dose Escalation Phase or starting Cycle 1 of the Dose Confirmation Phase. Pembrolizumab is administered IV at PDL2 on Day 1 of each cycle for the Efficacy Expansion Phase (Arm G).
  Other Names: Keytruda®
  Arms: Confirmation: DL 1 Quavonlimab Schedule 1 + Pembro (NSCLC): Arm A; Confirmation: DL 1 Quavonlimab Schedule 2 + Pembro (NSCLC): Arm B; Confirmation: DL 2 Quavonlimab Schedule 1 + Pembro (NSCLC): Arm E; Confirmation: DL 2 Quavonlimab Schedule 2 + Pembro (NSCLC): Arm C; Confirmation: DL 2 Quavonlimab Schedule 2 + Pembro (SCLC): Arm D; Escalation: DL 2 Quavonlimab + Pembro: Cohort 2; Escalation: DL 3 Quavonlimab + Pembro: Cohort 3; Escalation: Dose Level (DL) 1 Quavonlimab + Pembro: Cohort 1; Expansion: DL1 Quavonlimab Schedule 2+PDL2 Pembro Schedule 2: Arm F
Drug: Pembrolizumab/Quavonlimab — Pembrolizumab/Quavonlimab is a coformulated product composed of quavonlimab at DL1 in combination with pembrolizumab at dose level 2 (PDL2).
  Other Names: MK-1308A
  Arms: Coformulation Phase in China: Pembrolizumab/Quavonlimab Schedule 2: Arm K; Coformulation: Pembrolizumab/Quavonlimab Schedule 2: Arm I

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of escalating doses of quavonlimab when used in combination with pembrolizumab in participants with advanced solid tumors.

DETAILED DESCRIPTION:
After screening, participants will be assigned to the Dose Escalation, Dose Confirmation, Efficacy Expansion, or Coformulation Phase. The Dose Escalation Phase will evaluate available PK and safety data including dose limiting toxicities (DLTs). The Dose Confirmation Phase will gather additional safety, tolerability, PK, and preliminary efficacy data of quavonlimab in combination with pembrolizumab, and will include first-line advanced/metastatic non-small cell lung cancer (NSCLC) and second line (and beyond) advanced/metastatic small cell lung cancer (SCLC). The purpose of the Efficacy Expansion Phase is to gather preliminary anti-tumor efficacy data for quavonlimab in combination with pembrolizumab as well as for quavonlimab monotherapy in the specific target population of programmed cell death protein 1 (PD-1)/programmed cell death ligand 1 (PD-L1) refractory melanoma. The Coformulation Phase will evaluate the safety and PK of a coformulated product of pembrolizumab/quavonlimab (MK-1308A) in comparison to that of the single, co-administered products given at the same dose and schedule, and include participants with advanced solid tumors and participants from mainland China.

ELIGIBILITY:
Inclusion Criteria:

For Dose Escalation Phase:

* Have any histologically- or cytologically-confirmed advanced/metastatic solid tumor (except NSCLC for Cohorts 2 and 3) by pathology report and have received, been intolerant to, been ineligible for, or refused all treatment known to confer clinical benefit

For Dose Confirmation Phase NSCLC Arms (A, B, C, and E):

* Have newly diagnosed histologically or cytologically-confirmed stage IIIB/stage IV NSCLC. Epidermal growth factor receptor (EGFR)-and anaplastic lymphoma kinase (ALK) translocation-directed therapy is not indicated as primary therapy. Participant must not have received prior systemic treatment for advanced NSCLC or must have received previous neoadjuvant and adjuvant chemotherapies ≥6 months before dosing of study drug if prior systemic treatment was given for early stage disease

For Dose Confirmation Phase SCLC Arm (Arm D):

* Have histologically- or cytologically-confirmed metastatic (Stage III/IV) SCLC with progressive disease after ≥1 platinum-based chemotherapy regimen. Participants with platinum-sensitive disease are eligible
* Have measurable disease by RECIST 1.1 as assessed by the local site investigator/radiology
* Have Eastern Cooperative Oncology Group (ECOG) Performance Scale status of 0 or 1
* A female participant is eligible to participate if she is not pregnant or breastfeeding and at least 1 of the following conditions applies:
* Is not a woman of child bearing potential (WOCBP) OR
* Is a WOCBP and using a contraceptive method that is highly effective during the intervention period and for at least 120 days after the last dose of pembrolizumab or pembrolizumab/quavonlimab, whichever comes last
* Female participants of childbearing potential must have negative urine or serum pregnancy test within 24 hours for urine and within 72 hours for serum prior to receiving the first dose of study treatment
* Male participants with a female partner(s) of child-bearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication and refrain from donating sperm during this period
* Must submit an evaluable baseline tumor sample for analysis (either a recent or archival tumor sample)

For Efficacy Expansion Phase Arms F and G:

* Have histologically/cytologically-confirmed unresectable Stage III or Stage IV melanoma per American Joint Committee on Cancer (AJCC) staging system version 8, not amenable to local therapy
* Have at least 1 measurable lesion by CT or MRI per RECIST 1.1 by BICR. Cutaneous lesions and other superficial lesions are not considered measurable lesions for the purposes of this protocol, but may be considered as non-target lesions
* Participants with unresectable Stage III or IV disease must have progressed on treatment with an anti-PD-1/L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies (combinations with anti-cytotoxic T-lymphocyte associated protein 4 [CTLA-4] agents will not be allowed)
* Participants who receive anti-PD-1 therapy as adjuvant treatment following complete resection of Stage III or IV melanoma and have disease recurrence (unresectable loco-regional disease or distant metastases) while on active treatment or within 6 months of stopping anti-PD-1 are eligible
* Have submitted pre-trial imaging and provided a baseline tumor sample
* Proto-oncogene B-raf (BRAF) V600 mutation-positive melanoma participants should have received targeted therapy for advanced or metastatic disease (eg, BRAF/MEK inhibitor, alone or in combination) prior to enrolling on this study; however, they are not required to progress on this treatment prior to enrollment
* BRAF V600E mutation-positive melanoma participants who have NOT received a BRAF inhibitor (either as adjuvant therapy or in the metastatic disease setting) with lactate dehydrogenase (LDH) < local upper limit of normal (ULN), no clinically significant tumor-related symptoms, and absence of rapidly progressing metastatic melanoma. Approximately 10 participants each from Arms F and G will have 2 mandatory biopsies

For Dose Coformulation Phase Arm I:

* Have any histologically- or cytologically-confirmed advanced/metastatic solid tumor by pathology report and have received, been intolerant to, been ineligible for or refused all treatment known to confer clinical benefit
* Meet all requirements for Dose Escalation Phase and Dose Confirmation Phase

For the Coformulation Phase - Arm K (China only):

* Have any histologically- or cytologically-confirmed advanced/metastatic solid tumor by pathology report and have received, been intolerant to, been ineligible for, or refused all treatment known to confer clinical benefit
* Be a Chinese participant residing in China.

Exclusion Criteria:

* For all phases of the study: Has received previous treatment with another agent targeting cytotoxic T lymphocyte leukocyte antigen (CTLA)-4

For Dose Confirmation Phase:

* Has received previous treatment with another agent targeting programmed cell death protein 1 (PD-1), programmed cell death ligand 1 (PD-L1), or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) prior to the first dose of study therapy, or has not recovered to Common Toxicity Criteria for Adverse Events (CTCAE) Grade 1 or better from any AEs that were due to cancer therapeutics administered more than 4 weeks earlier
* Has received lung radiation therapy of >30 Gray (Gy) within 6 months before the first dose of study treatment
* Is currently participating and receiving study therapy in a study of an investigational agent or has participated and received study therapy in a study of an investigational agent or has used an investigational device within 28 days of administration of quavonlimab.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 3 years

For Dose Escalation Cohorts (1-3) and Dose Confirmation Arms (A-E):

* Has known untreated central nervous system (CNS) metastases. Has known carcinomatous meningitis
* Has received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse events (irAE)
* Has had a severe hypersensitivity reaction to treatment with any monoclonal antibody or components of the study drug
* Has any active infection requiring therapy
* Has a history of interstitial lung disease, history of noninfectious pneumonitis that required steroids (or has current pneumonitis), or history of inflammatory bowel disease
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has clinically significant cardiac disease
* Has received a live or live attenuated vaccine within 28 days of planned treatment start
* Has known history of human immunodeficiency virus (HIV) and/or known active Hepatitis B or C infections, and/or known to be positive for hepatitis B surface antigen (HBsAg)/ hepatitis B virus (HBV) DNA
* Has known psychiatric or substance abuse disorders that would interfere with the participant's ability to cooperate with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with screening and for up to 120 days following cessation of pembrolizumab or pembrolizumab/quavonlimab
* Has not fully recovered from any effects of major surgery without significant detectable infection

For Arm F and G (Efficacy Expansion Phase) and Arm K (Coformulation Phase) ONLY:

* Has known active CNS metastases and/or carcinomatous meningitis
* Has not had resolution of anti-PD-1 antibody-related AEs, including immune-mediated AEs back to Grade ≤1 or baseline (not applicable to Arm K)
* Has not discontinued steroid treatment for an irAE for at least 2 weeks prior to the first dose of study drug (not applicable to Arm K)
* Has ocular melanoma (not applicable to Arm K)
* Has mucosal melanoma (not applicable to Arm K)
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (53):
- United States (5):
  - Banner MD Anderson Cancer Center ( Site 0013), Gilbert, Arizona
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0005), Hackensack, New Jersey
  - Tennessee Oncology Nashville ( Site 0004), Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, LLC (START) ( Site 0001), San Antonio, Texas
  - Inova Schar Cancer Institute ( Site 1001), Fairfax, Virginia
- Australia (8):
  - Blacktown Hospital. Western Sydney local health district ( Site 0009), Blacktown, New South Wales
  - Calvary Mater Newcastle ( Site 0025), Waratah, New South Wales
  - Melanoma Institute Australia ( Site 0017), Wollstonecraft, New South Wales
  - Gallipoli Medical Research Foundation-GMRF CTU ( Site 0019), Brisbane, Queensland
  - Cairns and Hinterland Hospital and Health Service ( Site 0020), Cairns, Queensland
  - Ashford Cancer Centre Research ( Site 0012), Kurralta Park, South Australia
  - Ballarat Health Services ( Site 0022), Ballarat, Victoria
  - Alfred Health ( Site 0018), Melbourne, Victoria
- Canada (5):
  - Sunnybrook Research Institute ( Site 1103), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 1104), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 1102), Montreal, Quebec
  - Jewish General Hospital ( Site 1105), Montreal, Quebec
  - McGill University Health Centre ( Site 1101), Montreal, Quebec
- Fundacion Arturo Lopez Perez ( Site 5601), Santiago, Region M. de Santiago, Chile
- China (3):
  - Beijing Cancer hospital-Digestive Oncology ( Site 5001), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital-Phase 1 Unite ( Site 5004), Chongqing, Chongqing Municipality
  - Sir Run Run Shaw Hospital-Medical Oncology ( Site 5003), Hangzhou, Zhejiang
- France (5):
  - Hopital La Timone ( Site 3303), Marseille, Bouches-du-Rhone
  - Institut Bergonie ( Site 3306), Bordeaux, Gironde
  - CHRU Lille - Hopital Claude Huriez ( Site 3302), Lille, Nord
  - CH Lyon Sud Hospices Civils de Lyon ( Site 3307), Pierre-Bénite, Rhone
  - Gustave Roussy ( Site 3305), Villejuif, Val-de-Marne
- Regional General Hospital of Athens "Laiko" ( Site 3001), Athens, Attica, Greece
- Israel (3):
  - Rambam Medical Center ( Site 0003), Haifa
  - Hadassah Ein Karem Hebrew University Medical Center ( Site 0021), Jerusalem
  - Sheba Medical Center - Cancer Center ( Site 0002), Ramat Gan
- Italy (3):
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 3903), Napoli
  - IRCCS Istituto Oncologico Veneto ( Site 3905), Padua
  - Policlinico Le Scotte - A.O. Senese ( Site 3907), Siena
- Japan (2):
  - National Cancer Center Hospital East ( Site 0014), Kashiwa, Chiba
  - Hyogo Cancer Center ( Site 0015), Akashi, Hyōgo
- New Zealand (2):
  - Canterbury District Health Board ( Site 0023), Christchurch, Canterbury
  - Auckland City Hospital ( Site 0016), Auckland
- Poland (2):
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwers Medyczn ( Site 4803), Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Oddzial Badan Wczesnych Faz ( Site 4801, Warsaw, Masovian Voivodeship
- South Africa (3):
  - Sandton Oncology Medical Group PTY LTD ( Site 2701), Johannesburg, Gauteng
  - Cape Town Oncology Trials Pty Ltd ( Site 2704), Kraaifontein, Western Cape
  - Cancercare Rondebosch Oncology ( Site 2706), Rondebosch, Western Cape
- South Korea (4):
  - Asan Medical Center ( Site 0006), Seoul, Seoul
  - Seoul National University Hospital ( Site 0007), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0008), Seoul
  - Samsung Medical Center ( Site 0010), Seoul
- Spain (5):
  - Instituto Catalan de Oncologia ICO - Hospital Duran i Reynals ( Site 3403), L'Hospitalet de Llobregat, Barcelona
  - Onkologikoa - Instituto Oncologico de San Sebastian ( Site 3405), Donostia / San Sebastian, Gipuzkoa
  - Hospital General Universitario de Valencia ( Site 3404), Valencia, Valenciana, Comunitat
  - Hospital Clinic i Provincial de Barcelona ( Site 3401), Barcelona
  - Hospital Universitario Virgen de la Macarena ( Site 3402), Seville
- Skanes Universitetssjukhus Lund. ( Site 4601), Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Perets R, Bar J, Rasco DW, Ahn MJ, Yoh K, Kim DW, Nagrial A, Satouchi M, Lee DH, Spigel DR, Kotasek D, Gutierrez M, Niu J, Siddiqi S, Li X, Cyrus J, Chackerian A, Chain A, Altura RA, Cho BC. Safety and efficacy of quavonlimab, a novel anti-CTLA-4 antibody (MK-1308), in combination with pembrolizumab in first-line advanced non-small-cell lung cancer. Ann Oncol. 2021 Mar;32(3):395-403. doi: 10.1016/j.annonc.2020.11.020. Epub 2020 Dec 2. PMID 33276076
- [Result] Cho BC, Yoh K, Perets R, Nagrial A, Spigel DR, Gutierrez M, Kim DW, Kotasek D, Rasco D, Niu J, Satouchi M, Ahn MJ, Lee DH, Maurice-Dror C, Siddiqi S, Ren Y, Altura RA, Bar J. Anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody quavonlimab in combination with pembrolizumab: Safety and efficacy from a phase I study in previously treated extensive-stage small cell lung cancer. Lung Cancer. 2021 Sep;159:162-170. doi: 10.1016/j.lungcan.2021.07.009. Epub 2021 Jul 18. PMID 34371366
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, twenty-one participants who progressed by radiographic evaluation on monotherapy with MK-1308 (Arm G) after consultation with the sponsor crossed over to the combination treatment arm (MK-1308 25 mg + Pembrolizumab 400 mg)
Groups:
- Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W: On cycle 1, day 1 of the dose escalation phase, participants with advanced solid tumors received 25 mg quavonlimab (MK-1308) monotherapy followed by 25 mg quavonlimab in combination with 200 mg pembrolizumab (pembro) every 3 weeks (Q3W) for cycles 2-5. Participants then received 200 mg pembrolizumab monotherapy Q3W starting on Cycle 6, for up to 35 cycles total (up to approximately 24 months).
- Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W: On cycle 1, day 1 of the dose escalation phase, participants with advanced solid tumor except non-small cell lung cancer (NSCLC) received 75 mg quavonlimab monotherapy followed by 75 mg quavonlimab in combination with 200 mg pembrolizumab Q3W for cycles 2-5. Participants then received 200 mg pembrolizumab monotherapy Q3W starting on Cycle 6, for up to 35 cycles total (up to approximately 24 months).
- Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W: On cycle 1, day 1 of the dose escalation phase, participants with advanced solid tumor except non-small cell lung cancer (NSCLC) received 200 mg quavonlimab monotherapy followed by 200 mg quavonlimab in combination with 200 mg pembrolizumab Q3W for cycles 2-5. Participants then received 200 mg pembrolizumab monotherapy Q3W starting on Cycle 6, for up to 35 cycles total (up to approximately 24 months).
- Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W: On cycle 1, day 1 of the dose confirmation phase and during all subsequent cycles, participants with advanced/metastatic NSCLC received 25 mg quavonlimab in combination with 200 mg pembrolizumab Q3W. Participants were treated for 35 cycles total (up to approximately 24 months).
- Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W: On cycle 1, day 1 of the dose confirmation phase, participants with advanced/metastatic NSCLC received 25 mg quavonlimab in combination with 200 mg pembrolizumab Q3W. On all subsequent cycles, participants received 200 mg pembrolizumab Q3W and 25 mg quavonlimab every 6 weeks (Q6W). Participants were treated for up to 35 cycles total (up to approximately 24 months).
- Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W: On cycle 1, day 1 of the dose confirmation phase, participants with advanced/metastatic NSCLC received 75 mg quavonlimab in combination with 200 mg pembrolizumab Q3W. On all subsequent cycles, participants received 200 mg pembrolizumab Q3W and 75 mg quavonlimab Q6W. Participants were treated for 35 cycles total (up to approximately 24 months).
- Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W: On cycle 1, day 1 of the dose confirmation phase, participants with advanced/metastatic small cell lung cancer (SCLC) received 75 mg quavonlimab in combination with 200 mg pembrolizumab Q3W. On all subsequent cycles, participants received 200 mg pembrolizumab Q3W and 75 mg quavonlimab Q6W. Participants were treated for 35 cycles total (up to approximately 24 months).
- Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W: On cycle 1, day 1 of the dose confirmation phase and during all subsequent cycles, participants with NSCLC received 75 mg quavonlimab in combination with 200 mg pembrolizumab Q3W. Participants were treated for 35 cycles total (up to approximately 24 months).
- Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin: On cycle 1, day 1 of the efficacy expansion phase and during all subsequent cycles, participants with programmed cell death protein 1 (PD-1)/programmed cell death ligand 1 (PD-L1) refractory melanoma received 25 mg quavonlimab in combination with 400 mg pembrolizumab. Both quavonlimab and pembrolizumab were administered Q6W for 24 months.
- Arm G: MK-1308 25 mg Q6W: On cycle 1, day 1 of the efficacy expansion phase and during all subsequent cycles, participants with PD-1/PD-L1 refractory melanoma received 25 mg quavonlimab Q6W for up to 24 months.
- Arm I: MK-1308A Q6W (Co-form): On cycle 1, day 1 of the coformulation (Co-form) phase and during all subsequent cycles, participants with advanced/metastatic solid tumors received 400 mg pembrolizumab co-formulated with 25 mg quavonlimab (MK-1308A) Q6W for 24 months.
- Arm K: MK-1308A Q6W (Co-form): On cycle 1, day 1 of the coformulation phase and during all subsequent cycles, participants in mainland China with advanced/metastatic solid tumors received 400 mg pembrolizumab co-formulated with 25 mg quavonlimab (MK-1308A) Q6W for 24 months.
Period: Overall Study
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Started | 14 | 18 | 8 | 40 | 40 | 41 | 40 | 14 | 111 | 40 | 29 | 20
Treated | 14 | 17 | 8 | 40 | 40 | 40 | 40 | 14 | 111 | 40 | 29 | 20
Crossed Over to Combination Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 18 | 8 | 40 | 40 | 41 | 40 | 14 | 111 | 40 | 29 | 20
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 4 | 2 | 2 | 5 | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 1 | 3 | 9 | 7 | 2 | 4 | 23 | 6 | 7 | 5
Not completed — Randomized by Mistake without Study Treatment | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Death | 12 | 17 | 7 | 32 | 29 | 30 | 33 | 9 | 84 | 33 | 22 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form) | Total
Number analyzed (Participants) | 14 | 18 | 8 | 40 | 40 | 41 | 40 | 14 | 111 | 40 | 29 | 20 | 415
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 2 | 23 | 18 | 17 | 17 | 4 | 53 | 24 | 16 | 14 | 208
  >=65 years | 6 | 6 | 6 | 17 | 22 | 24 | 23 | 10 | 58 | 16 | 13 | 6 | 207
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 4 | 10 | 12 | 17 | 16 | 5 | 34 | 18 | 13 | 8 | 158
  Male | 3 | 8 | 4 | 30 | 28 | 24 | 24 | 9 | 77 | 22 | 16 | 12 | 257
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 11
  Not Hispanic or Latino | 13 | 17 | 7 | 40 | 37 | 41 | 39 | 13 | 102 | 33 | 29 | 20 | 391
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 8 | 3 | 0 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 30 | 26 | 26 | 16 | 8 | 3 | 0 | 3 | 20 | 132
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  White | 14 | 17 | 8 | 10 | 14 | 14 | 23 | 6 | 105 | 38 | 23 | 0 | 272
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥1 Dose Limiting Toxicity (DLT)
Description: DLT was defined as toxicity that is possibly, probably, or definitely related to study therapy and may result in a change in the given dose. DLTs include Grade (Gr)4 non-hematologic toxicity (not laboratory); Gr 4 hematologic toxicity lasting ≥7 days (except thrombocytopenia); most non-hematologic AEs ≥ Gr 3 in severity; any Gr 3 or Gr 4 non-hematologic laboratory value that requires clinically significant medical intervention, leads to hospitalization, persists for >1 week, or results in a drug-induced liver injury; Gr 3 or Gr 4 febrile neutropenia; a prolonged delay in initiating Cycle 2 or 3 of Dose Escalation or Cycle 2 of Dose Confirmation due to treatment-related toxicity; any treatment-related toxicity that causes the participant to discontinue treatment during the DLT observation period, and Gr 5 toxicity.
Time Frame: Up to 6 weeks
Population: The DLT evaluable population consists of all participants who received ≥1 dose of study treatment who finished the DLT observation period in the dose escalation or dose confirmation phase. Per protocol, no analysis was planned for the efficacy expansion phase (Arms F and G), coformulation phase (Arms I and K) and cross over phase (MK-1308 25 mg and Pembrolizumab 400 mg).
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 13 | 15 | 7 | 40 | 40 | 40 | 40 | 14 | 0 | 0 | 0 | 0
Percentage of Participants | 0.0 [0.0 to 10.9] | 13.3 [4.9 to 26.6] | 0.0 [0.0 to 18.2] | 7.5 [3.3 to 14.0] | 5.0 [1.7 to 10.8] | 10.0 [5.0 to 17.1] | 10.0 [5.0 to 17.1] | 7.1 [1.4 to 19.4] |  |  |  |

2. Primary Outcome: Number of Participants With ≥1 Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment. Per protocol, no analysis was planned for the cross over phase. The number of participants who experienced an AE are presented.
Time Frame: Up to approximately 77 months
Population: All participants who received at least one dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 14 | 17 | 8 | 40 | 40 | 40 | 40 | 14 | 111 | 40 | 29 | 20
Participants | 14 | 17 | 8 | 39 | 38 | 40 | 38 | 14 | 104 | 37 | 28 | 18

3. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment. Per protocol, no analysis was planned for the cross over phase. The number of participants who discontinued study treatment due to an AE are presented.
Time Frame: Up to approximately 26 months
Population: All participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 14 | 17 | 8 | 40 | 40 | 40 | 40 | 14 | 111 | 40 | 29 | 20
Participants | 1 | 4 | 3 | 7 | 7 | 17 | 7 | 6 | 14 | 1 | 4 | 2

4. Primary Outcome: Efficacy Expansion: Objective Response Rate (ORR) as Assessed by Blinded Independent Central Review (BICR) Based on Adjusted Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per adjusted Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR in the concurrent randomized subset as assessed by Blinded Independent Central Review (BICR) will be presented. Per protocol, only data for arms F and G were presented for this endpoint.
Time Frame: Up to approximately 72 months
Population: All participants with a baseline scan that demonstrated measurable disease and who were administered at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Arm I: MK-1308A Q6W (Co-form): On cycle 1, day 1 of the coformulation (Co-form) phase and during all subsequent cycles, participants with advanced/metastatic solid tumors received 400 mg pembrolizumab co-formulated with 25 mg quavonlimab (MK-1308A) for 24 months.
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 40 | 0 | 0
Percentage of participants |  |  |  |  |  |  |  |  | 4.9 [0.6 to 16.5] | 2.5 [0.1 to 13.2] |  |
Statistical Analysis 1: Comparison: Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin vs Arm G: MK-1308 25 mg Q6W; Test type: Other; Percent Difference; Comparision based on Miettinen & Nurminen method; Percent Difference = 2.4, 95% CI 2-sided [-8.7 to 14.1]

5. Secondary Outcome: Area Under the Plasma Concentration Time Curve (AUC) of Pembrolizumab
Description: AUC was defined as a measure of pembrolizumab exposure that was calculated as the product of plasma drug concentration and time after drug administration. AUC determined by blood samples collected pre-dose and at designated timepoints post-dose are presented. Per protocol, no analysis was planned for participants in arm G and cross over phase. AUC of pembrolizumab is presented. Blood sampling was taken for Cohorts 1-3: Predose and Postdose on Days 1, 8, 15 on Cycles 2 and 3. Arms A, B, C, D, E: Predose and Postdose on Days 1, 8, 15 on Cycles 1, 2, 3. Arm F: Predose and Postdose on Day 1 and 21 on Cycles 1, 2, 3. Arm I: Predose and Postdose on Day 1 and 21 on Cycles 1, 2, 3. Arm K: Predose and Postdose on Days 1, 2, 8, 15, 21 on Cycles 1, 2; Days 1, 21 on Cycle 3. Each cycle is 21 days.
Time Frame: At designated time points up to - Cohorts 1-3: Day 15 Cycle 3, Arms A, B, C, D, E: Day 15 Cycle 3, Arm F: Day 21 Cycle 3, Arm I: Day 21 Cycle 3, Arm K: Day 21 Cycle 3. Each cycle is 21 days.
Population: Participants who complied with the protocol sufficiently to ensure that their data will be likely to show the effects of treatment, according to the underlying scientific model and had available data from at least 1 dose of study intervention.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 11 | 8 | 3 | 30 | 34 | 27 | 28 | 9 | 31 | 0 | 8 | 20
day*μg/mL
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 30 | 34 | 27 | 28 | 9 | 31 | 0 | 8 | 20
  Cycle 1 |  |  |  | 608 (24.6) | 620 (25.9) | 627 (20.6) | 642 (23.9) | 554 (15.6) | 2050 (33.6) |  | 2250 (18.7) | 1610 (25.0)
  Cycle 2: number analyzed (Participants) | 11 | 8 | 3 | 30 | 31 | 24 | 26 | 9 | 18 | 0 | 5 | 16
  Cycle 2 | 729 (18.3) | 546 (40.5) | 727 (24.5) | 788 (24.7) | 854 (19.9) | 822 (25.0) | 877 (28.3) | 794 (18.0) | 2370 (40.6) |  | 2820 (29.7) | 1770 (34.4)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 21 | 27 | 19 | 15 | 7 | 16 | 0 | 2 | 6
  Cycle 3 |  |  |  | 911 (22.7) | 971 (22.9) | 944 (26.0) | 1050 (20.8) | 872 (16.3) | 2410 (29.5) |  | 3410 (16.1) | 2440 (39.8)

6. Secondary Outcome: Maximum Concentration (Cmax) of Pembrolizumab
Description: Cmax was defined as the maximum concentration of pembrolizumab observed in plasma. Cmax determined by blood samples collected pre-dose and at designated timepoints post-dose are presented. Per protocol, no analysis was planned for participants in arm G and cross over phase. Cmax of pembrolizumab is presented. Blood sampling was taken for Cohorts 1-3: Predose and Postdose on Days 1, 8, 15 on Cycles 2 and 3. Arms A, B, C, D, E: Predose and Postdose on Days 1, 8, 15 on Cycles 1, 2, 3. Arm F: Predose and Postdose on Day 1 and 21 on Cycles 1, 2, 3. Arm I: Predose and Postdose on Day 1 and 21 on Cycles 1, 2, 3. Arm K: Predose and Postdose on Days 1, 2, 8, 15, 21 on Cycles 1, 2; Days 1, 21 on Cycle 3. Each cycle is 21 days.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 13 | 13 | 8 | 39 | 40 | 37 | 39 | 14 | 105 | 0 | 28 | 20
μg/mL
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 39 | 40 | 37 | 39 | 14 | 105 | 0 | 28 | 20
  Cycle 1 |  |  |  | 71.8 (24.0) | 77.1 (26.7) | 74.0 (27.8) | 73.6 (22.3) | 70.9 (35.3) | 149 (29.1) |  | 149 (23.8) | 128 (21.9)
  Cycle 2: number analyzed (Participants) | 13 | 13 | 8 | 34 | 33 | 30 | 31 | 10 | 94 | 0 | 21 | 16
  Cycle 2 | 79.8 (31.3) | 82.3 (32.3) | 78.7 (32.4) | 82.9 (20.2) | 88.2 (20.9) | 83.9 (23.2) | 90.4 (23.7) | 84.8 (18.6) | 150 (28.9) |  | 164 (22.8) | 139 (20.5)
  Cycle 3: number analyzed (Participants) | 10 | 11 | 3 | 31 | 32 | 28 | 26 | 8 | 63 | 0 | 13 | 12
  Cycle 3 | 93.9 (21.0) | 74.9 (28.1) | 88.6 (12.2) | 84.2 (16.9) | 92.3 (27.5) | 91.8 (21.7) | 98.0 (27.4) | 84.5 (13.8) | 153 (22.1) |  | 168 (22.3) | 138 (31.1)

7. Secondary Outcome: Minimum Concentration (Cmin) of Pembrolizumab
Description: Cmin was defined as the minimum or "trough" concentration of pembrolizumab observed after its administration and just prior to the administration of a subsequent dose. Cmin determined by blood samples collected pre-dose and at designated timepoints post-dose are presented. Per protocol, no analysis was planned for participants in arm G and cross over phase. Cmin of pembrolizumab is presented. Blood sampling was taken for Cohorts 1-3: Predose and Postdose on Days 1, 8, 15 on Cycles 2 and 3, Day 1 on Cycle 4. Arms A, B, C, D, E: Predose and Postdose on Days 1, 8, 15 on Cycles 1, 2, 3. Arm F: Predose and Postdose on Day 1 and 21 on Cycles 1, 2, 3. Arm I: Predose and Postdose on Day 1 and 21 on Cycles 1, 2, 3. Arm K: Predose and Postdose on Days 1, 2, 8, 15, 21 on Cycles 1, 2; Days 1, 21 on Cycle 3. Each cycle is 21 days.
Time Frame: At designated time points up to - Cohorts 1-3: Day 1 Cycle 4, Arms A, B, C, D, E: Day 15 Cycle 3, Arm F: Day 21 Cycle 3, Arm I: Day 21 Cycle 3, Arm K: Day 21 Cycle 3. Each cycle is 21 days.
Population: as for outcome 5
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 11 | 10 | 3 | 33 | 35 | 30 | 29 | 9 | 92 | 0 | 21 | 16
μg/mL
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 33 | 35 | 30 | 29 | 9 | 92 | 0 | 21 | 16
  Cycle 1 |  |  |  | 13.3 [0.00 to 22.3] | 13.1 [3.93 to 24.9] | 14.3 [5.59 to 90.4] | 15.6 [6.35 to 35.9] | 11.5 [4.77 to 18.0] | 21.9 [1.89 to 143] |  | 19.5 [7.25 to 35.8] | 14.4 [5.74 to 26.0]
  Cycle 2: number analyzed (Participants) | 11 | 10 | 3 | 31 | 33 | 28 | 28 | 9 | 63 | 0 | 13 | 12
  Cycle 2 | 18.3 [11.3 to 27.8] | 11.3 [0.00 to 28.1] | 19.0 [9.21 to 24.6] | 19.6 [6.62 to 37.4] | 24.3 [9.06 to 34.6] | 20.4 [9.19 to 44.9] | 25.2 [10.1 to 55.1] | 18.9 [8.52 to 25.5] | 23.1 [0.0266 to 51.6] |  | 30.0 [16.2 to 60.4] | 22.5 [8.74 to 37.1]
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 22 | 28 | 20 | 18 | 7 | 43 | 0 | 9 | 9
  Cycle 3 |  |  |  | 25.7 [13.7 to 40.3] | 27.5 [12.4 to 42.2] | 25.5 [11.3 to 98.2] | 29.3 [10.4 to 56.7] | 27.7 [14.5 to 30.5] | 24.5 [2.22 to 127] |  | 34.0 [18.9 to 72.2] | 26.6 [7.74 to 32.6]
  Cycle 4: number analyzed (Participants) | 4 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 4 | 34.3 [29.8 to 39.9] | 14.1 [0.00 to 38.1] | 23.5 [23.5 to 23.5] |  |  |  |  |  |  |  |  |

8. Secondary Outcome: Area Under the Plasma Concentration Time Curve (AUC) of Quavonlimab (MK-1308)
Description: AUC was defined as a measure of quavonlimab exposure that was calculated as the product of plasma drug concentration and time after drug administration. AUC determined by blood samples collected pre-dose and at designated timepoints post-dose are presented. Per protocol, no analysis was planned for the cross over phase. AUC of quavonlimab is presented. Blood sampling was taken for Cohorts 1-3: Predose and Postdose on Days 1, 8, 15 on Cycles 1, 2 and 3. Arms A, B, C, D, E: Days 1, 8, 15 on Cycles 1, 2, 3. Arms F, G and I: Predose and Postdose on Day 1 and 21 on Cycles 1, 2, 3. Arm K: Days 1, 2, 8, 15, 21 on Cycles 1, 2; Days 1, 21 on Cycle 3. Each cycle is 21 days.
Time Frame: At designated time points up to - Cohorts 1-3: Day 15 Cycle 3, Arms A, B, C, D, E: Day 15 Cycle 3, Arm F, G, I: Day 21 Cycle 3, Arm K: Day 21 Cycle 3. Each cycle is 21 days.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 10 | 13 | 8 | 26 | 21 | 28 | 28 | 10 | 34 | 9 | 8 | 20
day*μg/mL
  Cycle 1 | 68.2 (17.7) | 160 (19.5) | 510 (25.7) | 55.0 (26.6) | 69.6 (33.5) | 199 (36.2) | 222 (39.7) | 178 (17.6) | 77.1 (32.7) | 92.8 (38.1) | 106 (34.7) | 85.8 (24.2)
  Cycle 2: number analyzed (Participants) | 8 | 4 | 3 | 21 | 0 | 0 | 0 | 8 | 18 | 4 | 5 | 14
  Cycle 2 | 91.5 (19.9) | 178 (53.9) | 751 (23.4) | 73.6 (26.4) |  |  |  | 192 (17.7) | 94.4 (43.9) | 65.9 (27.8) | 96.1 (39.7) | 86.0 (47.7)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 16 | 20 | 19 | 16 | 6 | 17 | 3 | 2 | 6
  Cycle 3 |  |  |  | 64.3 (56.5) | 59.4 (74.9) | 182 (75.1) | 193 (90.8) | 186 (22.1) | 95.2 (63.4) | 95.0 (58.2) | 72.1 (9.92) | 92.3 (60.2)

9. Secondary Outcome: Maximum Concentration (Cmax) of Quavonlimab
Description: Cmax was defined as the maximum concentration of quavonlimab observed in plasma. Cmax determined by blood samples collected pre-dose and at designated timepoints post-dose are presented. Per protocol, no analysis was planned for the cross over phase. Cmax of quavonlimab is presented. Blood sampling was taken for Cohorts 1-3: Predose and Postdose on Days 1, 8, 15 on Cycles 1, 2 and 3. Arms A, B, C, D, E: Days 1, 8, 15 on Cycles 1, 2, 3. Arms F, G and I: Predose and Postdose on Day 1 and 21 on Cycles 1, 2, 3. Arm K: Days 1, 2, 8, 15, 21 on Cycles 1, 2; Days 1, 21 on Cycle 3. Each cycle is 21 days.
Time Frame: as for outcome 8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 13 | 17 | 8 | 38 | 39 | 38 | 38 | 14 | 106 | 37 | 27 | 20
μg/mL
  Cycle 1: number analyzed (Participants) | 12 | 17 | 8 | 38 | 39 | 38 | 38 | 14 | 106 | 37 | 27 | 20
  Cycle 1 | 8.23 (26.1) | 22.5 (29.8) | 68.3 (17.2) | 7.28 (30.6) | 8.02 (29.5) | 23.4 (24.3) | 24.1 (30.1) | 25.0 (20.6) | 7.25 (26.4) | 7.42 (30.4) | 8.06 (26.5) | 8.23 (26.7)
  Cycle 2: number analyzed (Participants) | 13 | 10 | 7 | 35 | 0 | 0 | 0 | 10 | 95 | 33 | 21 | 16
  Cycle 2 | 9.41 (20.4) | 23.5 (25.1) | 71.9 (29.0) | 8.58 (22.4) |  |  |  | 26.3 (24.7) | 7.65 (25.3) | 7.22 (29.3) | 8.17 (26.2) | 7.99 (29.7)
  Cycle 3: number analyzed (Participants) | 10 | 9 | 3 | 31 | 32 | 26 | 26 | 7 | 65 | 11 | 13 | 12
  Cycle 3 | 9.11 (24.7) | 23.3 (48.0) | 88.3 (16.0) | 7.72 (27.7) | 6.98 (43.7) | 22.7 (33.1) | 24.2 (50.4) | 27.2 (10.2) | 7.94 (29.6) | 6.65 (32.7) | 7.25 (21.9) | 7.94 (35.4)

10. Secondary Outcome: Minimum Concentration (Cmin) of Quavonlimab
Description: Cmin was defined as the minimum or "trough" concentration of quavonlimab observed after its administration and just prior to the administration of a subsequent dose. Cmin determined by blood samples collected pre-dose and at designated timepoints post-dose are presented. Per protocol, no analysis was planned for the cross over phase. Cmin of quavonlimab is presented. Blood sampling was taken for Cohorts 1-3: Predose and Postdose on Days 1, 8, 15 on Cycles 1, 2 and 3. Arms A, B, C, D, E: Days 1, 8, 15 on Cycles 1, 2, 3. Arms F, G and I: Predose and Postdose on Day 1 and 21 on Cycles 1, 2, 3. Arm K: Days 1, 2, 8, 15, 21 on Cycles 1, 2; Days 1, 21 on Cycle 3. Each cycle is 21 days.
Time Frame: as for outcome 8
Population: as for outcome 5
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 13 | 14 | 8 | 35 | 33 | 26 | 29 | 10 | 95 | 32 | 21 | 16
μg/mL
  Cycle 1 | 1.44 [0.00 to 2.11] | 3.29 [0.00 to 6.86] | 8.01 [1.51 to 17.8] | 1.05 [0.00 to 1.80] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 3.44] | 15.6 [6.35 to 35.9] | 3.20 [0.00 to 5.26] | 0.00 [0.00 to 1.65] | 0.00 [0.00 to 1.26] | 0.00 [0.00 to 2.02] | 0.00 [0.00 to 1.32]
  Cycle 2: number analyzed (Participants) | 11 | 10 | 3 | 31 | 0 | 0 | 28 | 8 | 62 | 11 | 13 | 12
  Cycle 2 | 1.75 [0.00 to 3.10] | 2.83 [0.00 to 10.3] | 17.4 [1.73 to 19.2] | 1.17 [0.00 to 2.73] |  |  | 25.2 [10.1 to 55.1] | 3.40 [1.35 to 6.32] | 0.00 [0.00 to 8.23] | 0.00 [0.00 to 2.09] | 0.00 [0.00 to 1.68] | 0.00 [0.00 to 1.65]
  Cycle 3: number analyzed (Participants) | 0 | 1 | 0 | 22 | 25 | 21 | 18 | 6 | 43 | 8 | 9 | 9
  Cycle 3 |  | 1.91 [1.91 to 1.91] |  | 1.42 [0.00 to 2.86] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 3.10] | 29.3 [10.4 to 56.7] | 2.91 [2.21 to 5.77] | 0.00 [0.00 to 7.50] | 0.00 [0.00 to 7.20] | 0.00 [0.00 to 2.37] | 0.00 [0.00 to 1.05]

11. Secondary Outcome: Number of Participants With Pembrolizumab Anti-drug Antibodies (ADAs)
Description: Non-Treatment emergent (TE) ADA refers to presence of ADAs (as determined by assay) in the absence of treatment with pembrolizumab (i.e., at predose). Evaluable participants (used as the denominator for analysis) are the total number of negative, inconclusive, and positive participants (non-treatment emergent, treatment emergent and treatment boosted). Inconclusive participants are the number of participants with no positive ADA samples present and the drug concentration in the last sample above the drug tolerance level. ADA determined by blood samples collected pre-dose and at designated timepoints post-dose are presented. Per protocol, no analysis was planned for arm G and cross over phase.
Time Frame: Cohorts 1-3: Predose and day 1 of cycles 2, 3, 5, 6, 7, 9 and every 4 cycles up to 35 cycles. Arms A-E: Predose and day 1 of cycles 1-5, 6, 8 and every 4 cycles up to 35 cycles. Arms F, I, K: Predose and day 1 of cycles 1, 2, 3, 4. Each cycle is 21 days.
Population: Participants with at least one ADA sample available after treatment with pembrolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 12 | 13 | 5 | 36 | 39 | 37 | 35 | 11 | 103 | 0 | 23 | 20
Participants
  Evaluable | 12 | 13 | 5 | 36 | 39 | 37 | 35 | 11 | 103 |  | 23 | 20
  Negative | 12 | 12 | 5 | 31 | 33 | 33 | 31 | 10 | 94 |  | 20 | 13
  Non - TE Neutralizing Antibody (NAB) NEG (Negative): number analyzed (Participants) | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0
  Non - TE Neutralizing Antibody (NAB) NEG (Negative) |  | 1 |  |  |  |  |  |  |  |  | 1 |
  TE NAB NEG: number analyzed (Participants) | 0 | 0 | 0 | 36 | 39 | 37 | 35 | 11 | 103 | 0 | 0 | 20
  TE NAB NEG |  |  |  | 4 | 4 | 3 | 4 | 1 | 3 |  |  | 2
  TE NAB Positive (POS): number analyzed (Participants) | 0 | 0 | 0 | 36 | 0 | 37 | 0 | 0 | 0 | 0 | 0 | 20
  TE NAB Positive (POS) |  |  |  | 1 |  | 1 |  |  |  |  |  | 1
  Inconclusive: number analyzed (Participants) | 0 | 0 | 0 | 0 | 39 | 0 | 0 | 0 | 103 | 0 | 23 | 20
  Inconclusive |  |  |  |  | 2 |  |  |  | 5 |  | 2 | 4
  Treatment Boosted (TB) NAB NEG: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 103 | 0 | 0 | 20
  Treatment Boosted (TB) NAB NEG |  |  |  |  |  |  |  |  | 1 |  |  | 0

12. Secondary Outcome: Number of Participants With Quavonlimab Anti-drug Antibodies (ADAs)
Description: Non-Treatment emergent (TE) ADA refers to presence of ADAs (as determined by assay) in the absence of treatment with quavonlimab (i.e., at predose). Evaluable participants (used as the denominator for analysis) are the total number of negative, inconclusive, and positive participants (non-treatment emergent, treatment emergent and treatment boosted (TB)). Inconclusive participants are the number of participants with no positive ADA samples present and the drug concentration in the last sample above the drug tolerance level. ADA determined by blood samples collected pre-dose and at designated timepoints post-dose are presented. Per protocol, no analysis was planned for the cross over phase.
Time Frame: Cohort 1-3: Predose and day 1 of cycles 2, 3, 5, 6, 7, 9 and every 4 cycles up to 35 cycles. Arms A-E: Predose and day 1 of cycle 1-5, 6, 8 and every 4 cycles up to 35 cycles. Arms F, G, I, K: Predose and day 1 of cycles 1, 2, 3, 4. Each cycle is 21 days.
Population: Participants with at least one ADA sample available after treatment with quavonlimab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 14 | 15 | 8 | 36 | 39 | 37 | 35 | 11 | 102 | 38 | 23 | 20
Participants
  Evaluable | 14 | 15 | 8 | 36 | 39 | 37 | 35 | 11 | 102 | 38 | 23 | 20
  Negative | 3 | 7 | 4 | 12 | 6 | 6 | 8 | 4 | 35 | 21 | 8 | 6
  Non - Treatment Emergent Neutralizing Antibody (NAB) NEG (Negative): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TE NAB NEG: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TE NAB POS: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Inconclusive: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 102 | 38 | 0 | 20
  Inconclusive |  |  |  |  |  |  | 1 |  | 2 | 1 |  | 1
  TB NAB NEG: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TB NAB MISSING: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 37 | 0 | 0 | 102 | 38 | 0 | 20
  TB NAB MISSING |  | 1 |  |  |  | 1 |  |  | 3 | 2 |  | 2
  TE NAB MISSING | 11 | 7 | 4 | 23 | 32 | 30 | 26 | 7 | 61 | 13 | 15 | 11
  NON-TE NAB MISSING: number analyzed (Participants) | 0 | 0 | 0 | 36 | 39 | 0 | 0 | 0 | 102 | 38 | 0 | 0
  NON-TE NAB MISSING |  |  |  | 1 | 1 |  |  |  | 1 | 1 |  |

13. Secondary Outcome: Dose Escalation, Dose Confirmation, Coformulation: ORR as Assessed by Investigator Based on Adjusted RECIST v1.1
Description: ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented. Per protocol, no analysis was planned for the cross over phase.
Time Frame: Up to approximately 72 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 14 | 17 | 8 | 40 | 40 | 40 | 40 | 14 | 0 | 0 | 29 | 20
Percentage of participants | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 19.5] | 25.0 [3.2 to 65.1] | 32.5 [18.6 to 49.1] | 37.5 [22.7 to 54.2] | 30.0 [16.6 to 46.5] | 15.0 [5.7 to 29.8] | 35.7 [12.8 to 64.9] |  |  | 10.3 [2.2 to 27.4] | 20.0 [5.7 to 43.7]

14. Secondary Outcome: Efficacy Expansion: Duration of Response (DOR) as Assessed by BICR Based on Adjusted RECIST v1.1
Description: DOR was defined as the time from first documented evidence of complete response (CR: Disappearance of all target lesions) or confirmed partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by Blinded Independent Central Review (BICR) will be presented. Per protocol, only data for arms F and G were presented for this endpoint.
Time Frame: Up to approximately 72 months
Population: Participants who received at least one dose of study intervention who had either a CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 111 | 40 | 0 | 0
Months |  |  |  |  |  |  |  |  | NA [6.2 to NA] — NA = Median and lower limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 8.6 [8.6 to 8.6] |  |

ADVERSE EVENTS:
Time Frame: Up to approximately 77 months
Description: Analysis population for all-cause mortality consists of all allocated participants. Analysis population for safety consists of all participants who received at least one dose of study intervention.
Groups:
- Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin After Crossover: Participants who demonstrated radiographically confirmed progressive disease in Arm G and switched over to combination therapy received 25 mg quavonlimab in combination with 400 mg pembrolizumab. Both quavonlimab and pembrolizumab were administered Q6W for 24 months.
Arm/Group | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin After Crossover | Arm G: MK-1308 25 mg Q6W | Arm I: MK-1308A Q6W (Co-form) | Arm K: MK-1308A Q6W (Co-form)
All-Cause Mortality (participants affected / at risk) | 13/14 | 18/18 | 7/8 | 33/40 | 31/40 | 32/41 | 35/40 | 9/14 | 86/111 | 17/21 | 16/40 | 22/29 | 15/20
Serious Adverse Events (participants affected / at risk) | 2/14 | 10/17 | 4/8 | 20/40 | 14/40 | 23/40 | 16/40 | 10/14 | 31/111 | 4/21 | 9/40 | 15/29 | 4/20
Other Adverse Events (participants affected / at risk) | 14/14 | 16/17 | 8/8 | 38/40 | 38/40 | 38/40 | 37/40 | 13/14 | 102/111 | 17/21 | 31/40 | 26/29 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W (N=14) | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W (N=17) | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W (N=8) | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W (N=40) | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W (N=40) | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W (N=40) | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W (N=40) | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W (N=14) | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin (N=111) | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin After Crossover (N=21) | Arm G: MK-1308 25 mg Q6W (N=40) | Arm I: MK-1308A Q6W (Co-form) (N=29) | Arm K: MK-1308A Q6W (Co-form) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 9 (10) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W (N=14) | Cohort 2: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W (N=17) | Cohort 3: MK-1308 200 mg Q3W + Pembro. 200 mg Q3W (N=8) | Arm A: MK-1308 25 mg Q3W + Pembro. 200 mg Q3W (N=40) | Arm B: MK-1308 25 mg Q6W + Pembro. 200 mg Q3W (N=40) | Arm C: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W (N=40) | Arm D: MK-1308 75 mg Q6W + Pembro. 200 mg Q3W (N=40) | Arm E: MK-1308 75 mg Q3W + Pembro. 200 mg Q3W (N=14) | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin (N=111) | Arm F: MK-1308 25 mg Q6W + Pembro. 400 mg Q6W Co-admin After Crossover (N=21) | Arm G: MK-1308 25 mg Q6W (N=40) | Arm I: MK-1308A Q6W (Co-form) (N=29) | Arm K: MK-1308A Q6W (Co-form) (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 8 (9) | 5 (5) | 2 (3) | 11 (12) | 4 (4) | 8 (9) | 3 (4) | 5 (13)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 1 (1) | 3 (3) | 4 (4) | 3 (3) | 2 (2) | 7 (7) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 3 (3) | 0 (0) | 5 (5) | 9 (9) | 8 (8) | 8 (8) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 13 (13) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 3 (3) | 1 (1) | 4 (4) | 4 (4) | 5 (5) | 4 (4) | 3 (3) | 14 (17) | 2 (2) | 4 (4) | 4 (4) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2) | 3 (3) | 9 (18) | 3 (7) | 9 (15) | 10 (22) | 3 (6) | 27 (37) | 4 (4) | 3 (3) | 2 (4) | 3 (3)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 2 (2) | 9 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 10 (17) | 5 (5) | 2 (3) | 10 (16) | 0 (0) | 21 (24) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 5 (5) | 2 (2) | 5 (9) | 4 (4) | 3 (3) | 6 (6) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 2 (2) | 1 (3) | 4 (4) | 1 (1) | 13 (15) | 6 (6) | 4 (4) | 5 (5) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Early satiety (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (7) | 3 (3) | 2 (2) | 9 (13) | 9 (12) | 6 (8) | 11 (12) | 4 (5) | 26 (28) | 1 (1) | 6 (6) | 9 (9) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (7) | 1 (1) | 1 (1) | 1 (2) | 8 (12) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 4 (5) | 5 (10) | 3 (3) | 4 (7) | 9 (12) | 2 (2) | 2 (3) | 3 (3) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 5 (7) | 5 (6) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 2 (8) | 3 (3) | 0 (0) | 7 (8) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 10 (12) | 5 (5) | 9 (11) | 5 (7) | 6 (10) | 10 (13) | 1 (1) | 1 (1) | 2 (2) | 3 (4)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 3 (4) | 2 (2) | 9 (9) | 6 (6) | 11 (15) | 4 (6) | 6 (12) | 6 (9) | 3 (3) | 3 (3) | 3 (4) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 6 (6) | 4 (5) | 3 (3) | 2 (4) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood corticotrophin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 2 (4) | 2 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Cortisol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 3 (3) | 1 (1) | 4 (4) | 3 (4) | 4 (4) | 3 (3) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 5 (5) | 4 (4) | 3 (3) | 7 (7) | 4 (4) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 3 (3) | 13 (15) | 12 (13) | 8 (10) | 7 (8) | 1 (2) | 18 (19) | 2 (2) | 2 (2) | 2 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (10) | 2 (2) | 1 (1) | 3 (4) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (3) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 1 (1) | 2 (2) | 4 (9) | 5 (5) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 5 (7) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 3 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (3) | 4 (5) | 2 (2) | 1 (1) | 5 (10) | 2 (5) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 4 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 2 (2) | 2 (4) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 3 (5) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 1 (2) | 4 (4) | 6 (11) | 7 (11) | 4 (4) | 1 (1) | 14 (17) | 3 (3) | 3 (4) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 4 (4) | 2 (2) | 9 (9) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 5 (6) | 2 (2) | 0 (0) | 4 (4) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 9 (9) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 5 (7) | 2 (2) | 7 (7) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 7 (7) | 3 (3) | 5 (5) | 3 (3) | 2 (2) | 14 (15) | 3 (3) | 3 (4) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 5 (5) | 2 (2) | 2 (3) | 2 (3) | 8 (8) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 5 (7) | 5 (5) | 4 (4) | 6 (7) | 0 (0) | 10 (10) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 7 (7) | 7 (9) | 7 (7) | 5 (5) | 2 (2) | 9 (9) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (8) | 3 (4) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 5 (6) | 2 (2) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 6 (8) | 0 (0) | 12 (15) | 10 (15) | 11 (12) | 15 (20) | 5 (6) | 38 (42) | 2 (2) | 9 (9) | 11 (11) | 8 (10)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | 1 (1) | 11 (12) | 14 (16) | 13 (14) | 4 (6) | 6 (7) | 20 (25) | 0 (0) | 2 (2) | 8 (8) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3) | 0 (0) | 5 (5) | 3 (3) | 6 (10) | 8 (8) | 1 (6) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (12) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 5 (5) | 3 (4) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity was not directed by the Sponsor, the investigator agreed to submit all manuscripts or abstracts to the Sponsor before submission. This allowed the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT03179436/Prot_SAP_000.pdf